CLINICAL TRIAL: NCT04925258
Title: Supporting Parent and Child Engagement - SPACE Parenting Program
Brief Title: Supporting Parent and Child Engagement
Acronym: SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACE
Record Dates: First submitted 2021-05-03; First posted 2021-06-14 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2021-04

CONDITIONS: Stress, Psychological; Parenting; Covid19
MeSH Terms: conditions — Stress, Psychological; COVID-19

STUDY DESIGN:
Intervention Model Description: The study will recruit a group of parents and primary caregivers (e.g., mothers, fathers, adoptive parents, grandparents) who report elevated levels of parenting stress (above the 50th percentile of population norms on the Parenting Stress Index), and are the legal guardians of a child in the 3- to 4-year-old age range. Those parents will be randomly assigned to one treatment condition or the control condition. Parents in the treatment condition will participate in an 8-week parenting program that includes a combination of activities, parenting training, as well as drop-in sessions with a trained psychology student (MA-level or higher) or psychologist. The control group will receive services-as-usual (referral list for online and telehealth parenting and family mental health services).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Services-as-usual (No Intervention): Services-as-usual (referral list for online and telehealth parenting and family mental health services).
- SPACE Parenting Program (Experimental): The experimental groups of Manitoba-based parent-child dyads (children ages 3-4 years old) include:
  1. Weekly parenting materials, including online videos and mailed out parenting activities, that were developed for the Building Regulation in Dual Generations (BRIDGE) Therapy program. Also included are weekly drop-in group sessions with other parents facilitated by trained MA-level or higher psychology students or psychologists.
  Interventions: Behavioral: SPACE Parenting Program

INTERVENTIONS:
Behavioral: SPACE Parenting Program — The program involves a two-arm randomized trial of differing parenting interventions which include: a service as usual (SAU) cohort, in which parents are provided with local and online parenting and family mental health resources; An intervention group called SPACE that includes weekly parenting materials (i.e., two online ~10-minute videos, ten parent-child activities that were developed for the Building Regulation in Dual Generations (BRIDGE) Therapy program (NCT04347707 and NCT04639557) intervention group. Additionally, this group will receive weekly drop-in sessions with a facilitator-led (trained MA-level or higher psychology student or psychologist) interactive parenting group to re-enforce concepts and provide social support.
  Arms: SPACE Parenting Program

SUMMARY:
The COVID-19 pandemic and measures aimed at reducing the spread of the virus have created unique challenges and stresses for Canadian families. Balancing work, family, and daily life has become extremely difficult for many families. Economic uncertainty is widespread as many parents are dealing with increased demands such as working from home, running the household, and homeschooling and caring for their children without the support of their social networks. Recent findings from a study on the impact of the COVID-19 pandemic on young families conducted by our lab found that parents reported increased levels of stress, difficulties in following through with their parenting duties, and challenges managing their children's behaviour. Accessible programs are urgently needed to help parents cultivate supportive family relationships during and in recovery from the COVID-19 pandemic as physical distancing and public health requirements have further decreased the accessibility of existing programming. The proposed research aims to test the relative value of multiple light-touch parenting supports (developed through the REB-approved BRIDGE program, NCT04347707 and NCT04639557) in a 2-arm randomized control trial including behaviour management and emotion-focused strategies delivered through psychoeducational parenting videos, structured family activities, and an online parenting support group. The investigators plan to evaluate the efficacy of this program at reducing parenting stress (primary outcome) and promoting family well-being (secondary outcomes).

DETAILED DESCRIPTION:
Supportive parent-child relationships are increasingly understood to be the single most important predictor of resilient child development because they shape children's ability to build relationships and navigate the world around them. The emergence of emotion regulation skills during the preschool years serves as a key step in adaptive trajectories through which children learn to communicate their needs, engage in prosocial behaviour, and prepare for learning opportunities at school and beyond. Unfortunately, the COVID-19 pandemic has placed striking pressure on parents' capacities to engage in consistently supportive interactions due to factors such as limited childcare, financial strain, and poor mental health, which each present risks for child development.

The team of investigators designed the SPACE Program (Supporting Parent And Child Emotional well-being) to directly and immediately respond to family needs, with the potential for long-term impacts through its highly scalable approach. SPACE brings together best practices in emotion-focused parenting in a format guided by our Parent Advisory Board and over 1000 families who described their unmet needs in our rapid-response Parenting During the Pandemic survey. SPACE includes the provision of materials (i.e., psychoeducational videos and hands-on emotion-focused activities) alongside a virtual and interactive, facilitator-led parenting group to re-enforce skill acquisition and provide social support. The investigators' mixed-methods assessments are designed to understand the impacts of SPACE across multiple indicators of family function. The long-term goal is to create an accessible evidence-based online parenting program to promote child emotional development and well-being.

There are three objectives for the SPACE parenting project:

1. Assess the benefits of the novel SPACE program on parenting stress and parenting quality compared to services as usual (SAU): free provincial parenting resource guides and parenting sheets.
2. Determine the extent to which the SPACE program impacts child emotion-regulation development and if this relationship is mediated by parents' emotional and behavioural change.
3. Identify baseline factors linked to differential efficacy of SPACE. Hypothesis: SPACE will have higher efficacy for improving outcomes for children who a) identify as girls, b) exhibit higher cognitive performance, and c) exhibit greater cardiac flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Manitoba residence, parenting status (i.e., legal guardianship)
* Parents 18 years old or older
* Child/children's age group (ages 3-4)
* Elevated Parenting Stress Index- Short form (PSI-SF) scores (falling into the upper 50% range)
* English proficiency
* Access to a device with a camera (Smart phone, tablet, computer)

Exclusion Criteria:

* Resides outside Manitoba
* Parents under 18 years old
* Parents do have not legal guardianship of child
* Child <3 years or >4 years
* Parenting Stress Index- Short form (PSI-SF) score in bottom 50% range
* Not proficient in English
* No access to a device with a camera (Smart phone, tablet, computer)

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Change in parenting stress | : Time 1 prior to the beginning SPACE Program to ensure participants meet the inclusion criteria (upper 50th percentile on the PSI) and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx. 3 months after
  The Parenting Stress Index - Short Form (PSI) is a 36-item self-report measure completed by parents to measure stress level within the context of parenting. Participants respond to items on a 5-point Likert scale. Responses to each item in a sub-category are totaled to calculate three subcategory scores, which are summed to represent a total parenting stress score. Higher scores indicate higher levels of parenting stress. Normal scores fall within the 15th to 85th percentile, and scores above the 85th percentile represent clinically elevated levels of stress.

SECONDARY OUTCOMES:
Change in child mental health and behaviour | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Child behaviour from pre-intervention to post-intervention: Strengths and Difficulties Questionnaire (SDQ). A 25-item instrument developed to detect psychosocial problems in children aged 3-16 years. A value is given to each selection of "not true," somewhat true," and "certainly true." It measures five factors: emotional problems, conduct problems, hyperactivity/inattention problems, peer problems, and prosocial behaviour. All subscales include five items and range from 0-10. A total score can be summed from the first four factors; the total score ranges from 0-40, with higher scores indicating greater difficulties. Scores on the fifth factor of prosocial behaviour range from 0-10, with a lower score on this scale being less favourable.
Change in child behaviour | Time 1 prior to beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx. 3 months after Time 2).
  The Parent Daily Report will be used to assess parent-reported child behaviors in past 24 hours. This scale assess child behaviour and degree of parental stress through 12-items. These items are reported on a 3-point Likert scale from "did not occur" (0) to "occurred and stressful" (2). Higher scores on an item indicate more negative child behaviours and more stressful experiences.
Change in parent depressive symptoms | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  The Patient Health Questionnaire - 9 (PHQ-9) is a self-administered diagnostic instrument used to assess symptoms of major depressive disorder. The measure uses a 4-point Likert scale to assess the frequency of symptoms ranging from "not at all" to "nearly every day." A total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms. This measure will be completed by participants weekly throughout the intervention.
Change in parent anxiety symptoms | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Generalized Anxiety Disorder - 7 item scale (GAD-7) is a brief self-report measure to screen for generalized anxiety disorder. Scores range from 0-21, with higher scores indicating more severe anxiety.
Change in parent anger symptoms | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  The PROMIS Emotional Distress - Anger - Short-Form is a brief self-report measure used to assess the domain of anger. The items are measured on a 5-point Likert scale from "never" (1) to "always" (5). Total scores range from 5 to 25, with higher scores indicating more severe anger.
Change in emotion-focused parenting practices | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2)
  The Parenting Scale (PS) is a self-report measure of parenting style. The scale uses 30 items to assess various aspects of parenting/caregiving on a 7-point Likert scale. Scores are measured on a scale of 1-7 on each item, with 7 being less effective measures. The scale produces three subscale scores of Laxness (5-items), Overreactivity (5-items), and Verbosity (3-items), as well as a total score that includes all items. Scores are calculated by summing the items and dividing by the number of items to create a mean score; for example, the total score ranges from 1-7. Higher scores represent less effective parenting.
Change in parenting practices | Time 1: prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx. 3 months after Time 2).
  The Parenting Young Children (PARYC) scale is a self-report measure containing 21 questions designed to address parenting behaviors relevant to caring for young children. The scale includes three subscales: Supporting Positive Behavior, Setting Limits, and Proactive Parenting. Items are scored on a 5-point Likert scale from "never" (1) to "always" (5). Total scores can be calculated for each scale with higher scores indicating more positive parenting behaviors.
Change in mindful parenting practices intervention | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  The Mindfulness in Parenting Questionnaire (MIPQ) is a 61-item self-report measure of parenting mindfully. Items are scored on a 5-point Likert scale from "never" to "almost always." Raw summed scores can be converted using the MIPQ conversion table to standardized Rasch scores with a mean of 100 and standard deviation of 15, with higher scores indicating more mindfulness in parenting practices.
Changes in perceived parental/caregiver resilience from pre-intervention to post-intervention | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Connor Davidson Resilience Scale - 2 item (CD-RISC) measures resilience and the ability to bounce back after a tragedy, trauma, or stressful event. The measure includes two items scored on a 5-point Likert scale. Total scores range from 0 to 8, with higher scores indicating greater resilience.
Changes in parent/child screen time pre and post intervention | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Screen Time Questionnaire is a self-reported measure of screen time before and during COVID-19. The scale was created for the current study and contains a combination of open-ended and Likert scale questions. No cumulative score is used; instead, items will be evaluated individually. Higher scores on individual Likert scales generally indicate higher screen time use.
Changes in parental/caregiver spanking practices from pre to post intervention | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Parental Spanking will be assessed using a single-item assessing the frequency of spanking on a child's bottom, restricted to the age 2-5 years due to mandatory reporting guidelines for child maltreatment. Higher scores indicate greater frequency.
Changes in family resources measured from pre to post intervention | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Financial Strain will be assessed using a single-item created for a previous study. The item assess strain of managing unexpected expenses. Likert scores are reverse coded with the final score indicating greater financial strain.
Changes in recent stressful events from pre to post intervention | Time period: Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1), and Time 3 (approx.. 3 months after Time 2).
  Recent Stressful Experiences (RSE) is a self-report measure of recent family stressors and coping. This scale was adapted for the current study and contains a combination of open-ended and Likert scale questions. No cumulative score is used; instead, items will be evaluated individually. Higher scores on individual Likert scales assessing stressors indicate more stressors; higher scores on individual Likert scales assessing coping indicate greater resilience.

OTHER OUTCOMES:
Change in child cognitive function | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1).
  Child cognitive function will be assessed with behavioural regulation tasks. Specifically, children will participate in the child version of the Stroop task, in which they will be required to say the opposite in response to pictures of Day/Night images and Happy/Sad faces.
Change in child cardiac flexibility | Time 1 prior to the beginning SPACE Program and at Time 2 once again after the program is complete (approx. 8 weeks after Time 1).
  Cardiac flexibility will be measured with a downloadable app called "Heart Rate Plus" and heart rates for parent and child measured three and five times throughout baseline and post-intervention assessments, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie E Roos, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share data linked only to a de-identified number and without identifiable information (e.g., no videos, birthdates etc.), on online open science data repositories, such as osf.io).
Supporting Information: CSR
Time Frame: It would become available when the investigators publish the results of the study.
Access Criteria: Access will be based on the academic journal's level of access and requirements (e.g., subscription). Open access will be preferred at the time of journal selection, as possible, and preprint articles will be submitted online (e.g., psyarxiv) as possible based on journal requirements.

REFERENCES:
- [Background] Abidin, R. R. (2012). Parenting stress index (4th ed.). Lutz, FL: PAR.
- [Background] Cameron EE, Joyce KM, Delaquis CP, Reynolds K, Protudjer JLP, Roos LE. Maternal psychological distress & mental health service use during the COVID-19 pandemic. J Affect Disord. 2020 Nov 1;276:765-774. doi: 10.1016/j.jad.2020.07.081. Epub 2020 Jul 20. PMID 32736186
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] McCaffrey, S., Reitman, D., & Black, R. (2017). Mindfulness in Parenting Questionnaire (MIPQ): Development and validation of a measure of mindful parenting. Mindfulness, 8(1), 232-246.
- [Background] Mieloo C, Raat H, van Oort F, Bevaart F, Vogel I, Donker M, Jansen W. Validity and reliability of the strengths and difficulties questionnaire in 5-6 year olds: differences by gender or by parental education? PLoS One. 2012;7(5):e36805. doi: 10.1371/journal.pone.0036805. Epub 2012 May 18. PMID 22629332
- [Background] McDaniel, B. T., Everest, J., & White, C. (April 2018). Parent distraction with technology and its impact on parenting quality. Poster presentation: Illinois Council on Family Relations. Normal, IL.
- [Background] PROMIS Health Organization & PROMIS Cooperative Group. (2012). Level 2 - Anger - Adult: PROMIS Emotional Distress - Anger - Short Form. Evanston: IL
- [Background] Rideout, V. (2017). The Common Sense census: Media use by kids age zero to eight. San Francisco, CA: Common Sense Media
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Perrin EC, Leslie LK, Boat T. Parenting as Primary Prevention. JAMA Pediatr. 2016 Jul 1;170(7):637-8. doi: 10.1001/jamapediatrics.2016.0225. No abstract available. PMID 27182902
- [Background] Luthar SS, Eisenberg N. Resilient Adaptation Among At-Risk Children: Harnessing Science Toward Maximizing Salutary Environments. Child Dev. 2017 Mar;88(2):337-349. doi: 10.1111/cdev.12737. Epub 2017 Feb 1. PMID 28144962
- [Background] Blair C, Diamond A. Biological processes in prevention and intervention: the promotion of self-regulation as a means of preventing school failure. Dev Psychopathol. 2008 Summer;20(3):899-911. doi: 10.1017/S0954579408000436. PMID 18606037
- [Background] Dixon Jr, W. E., & Smith, P. H. (2000). Links between early temperament and language acquisition. Merrill-Palmer Quarterly (1982-), 417-440.
- [Background] Eisenberg N, Sadovsky A, Spinrad TL. Associations of emotion-related regulation with language skills, emotion knowledge, and academic outcomes. New Dir Child Adolesc Dev. 2005 Fall;(109):109-18. doi: 10.1002/cd.143. PMID 16342899
- [Background] Eisenberg N, Valiente C, Eggum ND. Self-Regulation and School Readiness. Early Educ Dev. 2010 Sep 1;21(5):681-698. doi: 10.1080/10409289.2010.497451. PMID 21234283
- [Background] Howard SJ, Williams KE. Early Self-Regulation, Early Self-Regulatory Change, and Their Longitudinal Relations to Adolescents' Academic, Health, and Mental Well-Being Outcomes. J Dev Behav Pediatr. 2018 Jul/Aug;39(6):489-496. doi: 10.1097/DBP.0000000000000578. PMID 29781830
- [Background] Williams, K. E., & Berthelsen, D. (2017). The development of prosocial behaviour in early childhood: Contributions of early parenting and self-regulation. International Journal of Early Childhood, 49(1), 73-94. https ://doi.org/10.1007/s1315 8-017-0185-5.
- [Background] Spinelli M, Lionetti F, Setti A, Fasolo M. Parenting Stress During the COVID-19 Outbreak: Socioeconomic and Environmental Risk Factors and Implications for Children Emotion Regulation. Fam Process. 2021 Jun;60(2):639-653. doi: 10.1111/famp.12601. Epub 2020 Sep 28. PMID 32985703
- [Background] Roos LE, Salisbury M, Penner-Goeke L, Cameron EE, Protudjer JLP, Giuliano R, Afifi TO, Reynolds K. Supporting families to protect child health: Parenting quality and household needs during the COVID-19 pandemic. PLoS One. 2021 May 24;16(5):e0251720. doi: 10.1371/journal.pone.0251720. eCollection 2021. PMID 34029311